CLINICAL TRIAL: NCT02393365
Title: Prevalence and Screening of Hepatitis C in Belgium in 2015
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Dr Luc Lasser, Head of Clinic, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUB-HCV screening
Record Dates: First submitted 2015-03-09; First posted 2015-03-19 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; HCV; screening
MeSH Terms: conditions — Hepatitis C | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HCV screening (Other): All patients admitted to the one day clinic for surgery and gastroenterology.
  Interventions: Other: Questionnaire; Procedure: HCV serology

INTERVENTIONS:
Other: Questionnaire — All patients admitted to the one day clinic for surgery and gastroenterology will be asked, after signing an informed consent, to fill in a questionnaire about HCV risk factors.
Procedure: HCV serology — In case of a pre-operative blood sample an HCV serology will also be done as part of a routine pre-operative screening.
  In patients where no pre-operative blood sample is done an additional consent will be asked to perform a blood sample for HCV serology. This qualifies the study as 'interventional' according to the Belgian legislation.

SUMMARY:
Hepatitis C is caused by the hepatitis C virus (HCV) that causes inflammation of the liver that can lead to diminished liver function or liver failure.

The number of chronically infected persons worldwide is estimated to be about 170 million that is 2.35% of the world population. Most people infected with the hepatitis C virus have no symptoms of the disease until the advanced stages of liver disease have occurred, which may take several years. The long-term impact of HCV infection is highly variable, from minimal changes to extensive fibrosis and cirrhosis with or without hepatocellular carcinoma (HCC).

Advanced liver disease (ALD) can lead to significant clinical and economic consequences, including liver transplantation. HCV can reduce life expectancy and impair quality of life. HCV-related complications as well as the highly debilitating effects on patients represent a significant item of expenditure for the National Health Service. Because of the latency of infection, numerous country-specific population analyses suggest that HCV will cause an increasing number of liver-related deaths despite the dramatic drop in incidence and prevalence. These deaths will be related to prevalent HCV infection especially during and after World War II through indiscreet and widespread treatment with intravenous injection using contaminated syringes, needles and remunerated blood donors. Eradicating HCV infection can prevent the complications of HCV-related liver and extrahepatic diseases, including liver necroinflammation, fibrosis, cirrhosis, HCC, and death.

Newly discovered hepatitis C virus (HCV) therapy with direct acting antiviral agents (DAA) like Simeprevir, sofosbuvir open a new chapter in the treatment of chronic hepatitis C. Those new treatment regimens promise oral dosing, higher SVR, shorter duration of treatment and fewer side effects. In a near future all patients should qualify for future all-oral therapies.

However recent analysis have shown that increasing efficacy of treatment alone will not be able to reduce the HCV disease burden. The largest reduction in HCV-related morbidity and mortality can be obtained when higher efficacy therapies is combined with increased diagnosis and treatment rate. With a treatment rate of 10% it is possible to achieve a > 90% decline in total infections by 2030. This would require a 3-5 fold increase in diagnosis and/or treatment for most countries.

The implementation of screening criteria for hepatitis C virus (HCV) such as targeting birth cohorts has potential effect on reducing the progression of hepatitis C virus (HCV) to advanced liver disease (ALD) and could avoid unnecessary high financial costs and preserve quality of life.

Robust data from public health surveillance, surveys of the general and risk populations are required to make decisions in allocating public health resources to diagnose, assess and treat HCV infection.

In Belgium no recent prevalence studies have been conducted. The most cited anti-HCV prevalence is 0.87% based on a study in the Flemish population published in 1997 but collected in 1994. In a French Belgian population there was an overall seroprevalence of 0.6%. However, the population under study was not representative for the whole French community, because the recruited subjects were significantly younger.

A survey among cirrhotic and hepatocellular patients in the French community revealed that 20% of cirrhosis and 47% of hepatocellular cancer were related to hepatitis C. The diagnosis rate of HCV in Belgium is estimated at 43%, signifying that more than 50% of HCV patients remains undiagnosed.

Several studies have already mentioned that aged population especially those born after Second World War are carriers of hepatitis C virus infection. Early detection of HCV infection and treating before progress to advanced liver disease (ALD) is an excellent opportunity to rationalize resource allocation and to improve patients' quality of life.

Recently birth cohort screening recommendations were developed in the United States. In Belgium, no formal screening strategy exists. However the Belgian association of the study of the liver (BASL) recommends targeted HCV screening for high-risk populations (including individuals with a blood transfusion or major medical event prior to 1 july 1990, intranasal or IDU and dialysis patients) in addition to nontargeted screening among pre-operative patients and pregnant women. A birth cohort analysis based on a model suggests a birth cohort between 1950 and 1975 in Belgium. This population should reflect 70% of the viremic population.

In this study, the investigators want to estimate the prevalence of hepatitis C in Belgium in 2014 and to confirm the proposed targeted birth cohort and other risk factors. These data could provide an efficient source of identifying newly diagnosed patients as part of a national screening strategy.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the one day clinic for surgery and gastroenterology.

Exclusion Criteria:

* none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Actual)
Dates: Start 2015-03-10 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
HCV risk factors questionnaire | up to one day after hospital admission
  All patients admitted to the one day clinic for surgery and gastroenterology will be asked, after signing an informed consent, to fill in a questionnaire regarding HCV risk factors (1 page). The collection of the questionnaires and the entering of the data into an electronic database will be done in an anonymous way.
Positive/Negative Hepatitis C serology | up to 10 days after hospital admission
  In case of a pre-operative blood sampling, an HCV detection test will be done on the serum as part of the routine pre-operative screening. The sample will be analyzed in the Hospital Laboratory according to the current belgian guidelines regarding hepatitis C virus detection. In patients where no pre-operative blood sample is done, an additional consent will be asked to take a blood sample for HCV detection. In case of a positive test result (positive HCV serology), patients will be contacted. Those patients will be proposed to contact their family doctor (GP) or a specialist of their choice in order to realize a classic work up and discuss therapeutic options if necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Lasser, MD, Principal Investigator — CHU Brugmann; Christophe Moreno, MD, Principal Investigator — Erasme; Thomas Serste, MD, Principal Investigator — CHU St Pierre; Peter Starkel, MD, Principal Investigator — UCL - St Luc
Locations (4):
- Belgium (4):
  - St Pierre Hospital, Brussels
  - CHU Brugmann, Brussels
  - Erasme, Brussels
  - UCL St Luc, Brussels

REFERENCES:
- [Background] Lavanchy D. Evolving epidemiology of hepatitis C virus. Clin Microbiol Infect. 2011 Feb;17(2):107-15. doi: 10.1111/j.1469-0691.2010.03432.x. PMID 21091831
- [Background] European Association for Study of Liver. EASL Clinical Practice Guidelines: management of hepatitis C virus infection. J Hepatol. 2014 Feb;60(2):392-420. doi: 10.1016/j.jhep.2013.11.003. Epub 2013 Dec 9. No abstract available. PMID 24331294
- [Background] Menzin J, White LA, Nichols C, Deniz B. The economic burden of advanced liver disease among patients with hepatitis C virus: a large state Medicaid perspective. BMC Health Serv Res. 2012 Dec 15;12:459. doi: 10.1186/1472-6963-12-459. PMID 23241078
- [Background] Wong JB. Hepatitis C: cost of illness and considerations for the economic evaluation of antiviral therapies. Pharmacoeconomics. 2006;24(7):661-72. doi: 10.2165/00019053-200624070-00005. PMID 16802842
- [Background] Ruggeri M, Coretti S, Gasbarrini A, Cicchetti A. Economic assessment of an anti-HCV screening program in Italy. Value Health. 2013 Sep-Oct;16(6):965-72. doi: 10.1016/j.jval.2013.07.005. PMID 24041346
- [Background] Yoshizawa H. Hepatocellular carcinoma associated with hepatitis C virus infection in Japan: projection to other countries in the foreseeable future. Oncology. 2002;62 Suppl 1:8-17. doi: 10.1159/000048270. PMID 11868791
- [Background] Wedemeyer H, Duberg AS, Buti M, Rosenberg WM, Frankova S, Esmat G, Ormeci N, Van Vlierberghe H, Gschwantler M, Akarca U, Aleman S, Balik I, Berg T, Bihl F, Bilodeau M, Blasco AJ, Brandao Mello CE, Bruggmann P, Calinas F, Calleja JL, Cheinquer H, Christensen PB, Clausen M, Coelho HS, Cornberg M, Cramp ME, Dore GJ, Doss W, El-Sayed MH, Ergor G, Estes C, Falconer K, Felix J, Ferraz ML, Ferreira PR, Garcia-Samaniego J, Gerstoft J, Giria JA, Goncales FL Jr, Guimaraes Pessoa M, Hezode C, Hindman SJ, Hofer H, Husa P, Idilman R, Kaberg M, Kaita KD, Kautz A, Kaymakoglu S, Krajden M, Krarup H, Laleman W, Lavanchy D, Lazaro P, Marinho RT, Marotta P, Mauss S, Mendes Correa MC, Moreno C, Mullhaupt B, Myers RP, Nemecek V, Ovrehus AL, Parkes J, Peltekian KM, Ramji A, Razavi H, Reis N, Roberts SK, Roudot-Thoraval F, Ryder SD, Sarmento-Castro R, Sarrazin C, Semela D, Sherman M, Shiha GE, Sperl J, Starkel P, Stauber RE, Thompson AJ, Urbanek P, Van Damme P, van Thiel I, Vandijck D, Vogel W, Waked I, Weis N, Wiegand J, Yosry A, Zekry A, Negro F, Sievert W, Gower E. Strategies to manage hepatitis C virus (HCV) disease burden. J Viral Hepat. 2014 May;21 Suppl 1:60-89. doi: 10.1111/jvh.12249. PMID 24713006
- [Background] McGarry LJ, Pawar VS, Panchmatia HR, Rubin JL, Davis GL, Younossi ZM, Capretta JC, O'Grady MJ, Weinstein MC. Economic model of a birth cohort screening program for hepatitis C virus. Hepatology. 2012 May;55(5):1344-55. doi: 10.1002/hep.25510. Epub 2012 Mar 18. PMID 22135116
- [Background] Van Damme P, Thyssen A, Van Loock F. Epidemiology of hepatitis C in Belgium: present and future. Acta Gastroenterol Belg. 2002 Apr-Jun;65(2):78-9. PMID 12148442
- [Background] Dore GJ, Ward J, Thursz M. Hepatitis C disease burden and strategies to manage the burden (Guest Editors Mark Thursz, Gregory Dore and John Ward). J Viral Hepat. 2014 May;21 Suppl 1:1-4. doi: 10.1111/jvh.12253. PMID 24713003
- [Background] McEwan P, Ward T, Yuan Y, Kim R, L'italien G. The impact of timing and prioritization on the cost-effectiveness of birth cohort testing and treatment for hepatitis C virus in the United States. Hepatology. 2013 Jul;58(1):54-64. doi: 10.1002/hep.26304. Epub 2013 May 27. PMID 23389841
- [Background] Smith BD, Morgan RL, Beckett GA, Falck-Ytter Y, Holtzman D, Teo CG, Jewett A, Baack B, Rein DB, Patel N, Alter M, Yartel A, Ward JW; Centers for Disease Control and Prevention. Recommendations for the identification of chronic hepatitis C virus infection among persons born during 1945-1965. MMWR Recomm Rep. 2012 Aug 17;61(RR-4):1-32. PMID 22895429
- [Background] Van Damme P, Laleman W, Starkel P, Van Vlierberghe H, Vandijck D, Hindman SJ, Razavi H, Moreno C. Hepatitis C epidemiology in Belgium. Acta Gastroenterol Belg. 2014 Jun;77(2):277-9. PMID 25090833